CLINICAL TRIAL: NCT06879379
Title: A Randomized, Multicenter Study Comparing Post-Transplant KPD Regimen Consolidation With No Consolidation in Newly Diagnosed Multiple Myeloma (NDMM) Transplant-eligible Patients
Brief Title: KPD Consolidation After ASCT in NDMM Patients
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Jin Lu, MD, Deputy Director of Department of Hematology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024PHB165-001-202501
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Multiple Myeloma, Newly Diagnosed
Keywords: consolidation
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- KPD consolidation (Experimental): KPD consolidation therapy for 2 cycles, followed by maintenance
  Interventions: Drug: KPD (carfilzomib, pomalidomide, and dexamethasone) consolidation
- No consolidation (No Intervention): Direct maintenance without consolidation.

INTERVENTIONS:
Drug: KPD (carfilzomib, pomalidomide, and dexamethasone) consolidation — After post-transplant randomization, patients will receive either KPD (carfilzomib, pomalidomide, and dexamethasone) consolidation then maintenance or no consolidation and maintenance.
  Arms: KPD consolidation

SUMMARY:
This study aims to evaluate the efficacy and safety of post-transplant consolidation therapy with the KPD regimen (carfilzomib, pomalidomide, and dexamethasone) versus no consolidation, followed by maintenance therapy, in patients with transplant-eligible newly diagnosed multiple myeloma (TE-NDMM). The primary goal is to compare minimal residual disease (MRD) negativity rates and overall treatment outcomes between the two groups.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is a malignancy characterized by abnormal proliferation of plasma cells, leading to organ damage and poor prognosis. Despite advances in treatment, including autologous stem cell transplantation (ASCT), the disease remains incurable for most patients. Post-transplant consolidation and maintenance therapies have emerged as critical strategies to deepen remission and prolong progression-free survival (PFS). However, the role of consolidation therapy remains debated. This study aims to clarify whether KPD consolidation therapy after ASCT provides additional benefits compared to direct maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Newly diagnosed MM eligible for transplantation.
* Received upfront triplet or quadraplet induction regimen.
* Received upfront ASCT after induction.
* ECOG score < 2.
* Adequate Organ Function Reserve:

  1. Alanine aminotransferase (ALT) / Aspartate aminotransferase (AST) ≤ 2.5 × UNL (upper limit of normal);
  2. Serum total bilirubin ≤ 1.5 × UNL. If the patient has congenitally high bilirubin, direct bilirubin must be ≤ 1.5 × UNL;
  3. Left ventricular ejection fraction (LVEF) ≥ 50% as diagnosed by echocardiography, with no clinically significant electrocardiogram (ECG) abnormalities;
  4. Basal oxygen saturation > 95% in room air;
* Women of childbearing age agree to use effective contraceptive measures during the period of using the study drug and within 3 months after the last administration of the study drug; and to use highly effective contraceptive measures for at least 1 year thereafter. Male participants with fertile partners must agree to use effective barrier contraception during the period of using the study drug and within 3 months after the last administration of the study drug;
* The participant is willing and able to comply with the study procedures and voluntarily signs the written informed consent form.

Exclusion Criteria:

* Patients with primary plasma cell leukemia or POEMs syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes);
* Patients diagnosed with primary amyloidosis, Waldenström's macroglobulinemia, monoclonal gammopathy of undetermined significance, or smoldering multiple myeloma;
* Patients with severe mental disorders, altered mental status, or a history of central nervous system (CNS) diseases such as epileptic seizures, cerebral vascular ischemia/ hemorrhage, dementia, cerebellar diseases, or any autoimmune diseases involving the CNS;
* Patients with a history of the following genetic diseases: Fanconi anemia, Shwachman-Diamond syndrome, Costello syndrome, or any other known bone marrow failure syndrome;
* Patients who underwent a diagnosis or treatment for another malignancy within 1 year prior to randomization, or had a previous diagnosis of another malignancy with evidence of residual disease (excluding patients with any type of non-melanoma skin cancer or completely resected carcinoma in situ);
* Patients with active infectious diseases, known human immunodeficiency virus (HIV) positivity, or active hepatitis B or C infection;
* Patients known to be allergic to any of the study drugs, their analogs, or any excipients of the study drugs in various formulations;
* Patients with concurrent or suspected central nervous system infiltration;
* Patients with drug use, medical, psychological, or social conditions that may interfere with the participant's ability to participate in the study or the assessment of study outcomes;
* Pregnant or lactating women;
* Any other conditions deemed by the investigator as unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Minimal residual disease (MRD) negativity rate prior to maintenance therapy | 36 months
  The primary endpoint of this study is to compare the minimal residual disease (MRD) negativity rate prior to maintenance therapy in transplant-eligible newly diagnosed multiple myeloma (NDMM) patients who receive KPD consolidation therapy versus those who do not receive consolidation therapy after triplet or quadraplet induction therapy and autologous stem cell transplantation (ASCT).
Overall Response Rate (ORR) | 36 months
  Compare the overall response rate (ORR) including the rates of stringent complete response (sCR), complete response (CR), very good partial response (VGPR) and partial response (PR), prior to maintenance therapy according to the IMWG (International Myeloma Working Group) assessment criteria, between the two treatment groups。

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 36 months
  Time interval from ASCT to disease progression or death.
Overall Survival (OS) | 36 months
  Time interval from ASCT to death

CONTACTS AND LOCATIONS:
Overall Officials: Jin Lu, M.D., Principal Investigator — Peking University People's Hospital
Locations (3):
- China (3):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Fuxing Hospital affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality